CLINICAL TRIAL: NCT01782053
Title: Communicating Smoking Risks Through Graphic Warning Labels
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Dan Romer, Director, Adolescent Communication Institute, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1R01CA157824-01A1 (NIH)
Record Dates: First submitted 2013-01-29; First posted 2013-02-01 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Lung Cancer; Heart Disease
MeSH Terms: conditions — Lung Neoplasms; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control condition (Experimental): Current packaging with warning on side replaced with one of 9 mandated warning statements
  Interventions: Behavioral: Control
- Text plus picture (Experimental): Revised packaging with half of front and back of pack showing FDA proposed warning including image.
  Interventions: Behavioral: Picture warning
- Picture plus additional warning text (Experimental): Same as text plus picture but containing additional text elaborating on the basis for the warning.
  Interventions: Behavioral: Picture warning

INTERVENTIONS:
Behavioral: Picture warning — Warning contains picture proposed for each text statement by FDA
  Arms: Picture plus additional warning text; Text plus picture
Behavioral: Control
  Arms: Control condition

SUMMARY:
Smoking is the largest preventable health risk in the U.S. The Family Smoking Prevention and Tobacco Control Act of 2010 mandated the placement of larger pictorial warnings on cigarette packs as well as nine new statements of smoking risks. This trial tests the effectiveness of the warnings proposed by the Food and Drug Administration by providing cigarettes with the proposed labels to 320 smokers across two sites (Philadelphia, PA and Columbus, OH). In addition, the trial tests the effects of different warning label components.

ELIGIBILITY:
Inclusion Criteria:

* smoke between 5 and 40 cigarettes per day and 100 in lifetime
* Not currently trying to quit
* between 18 and 65 years of age

Exclusion Criteria:

* smokes 120's or roll-your own or noncommercial cigarettes
* pregnant or breastfeeding
* history of substance abuse past 5 years
* more than 25 standard alcohol drinks per week
* use of other nicotine products, such as cigars, nicotine gum
* current treatment for copd, cancer, pulmonary disease, alcohol/drug dependence
* current treatment for a psychiatric condition
* physical/visual/mental impairment that prevents reading from a computer screen
* not US resident
* unable to read English
* English not main language
* other member of household in study
* friend who smokes in study
* unable to attend weekly appointments between 9 am and 6 pm Monday-Friday
* unable to use hand-held computer to enter daily mood ratings

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Intention to try to quit smoking in next 30 days | Assessed after 4 weeks of exposure to new labels

SECONDARY OUTCOMES:
Affective reactions toward cigarettes and smoking cues | After 4 weeks of exposure to the new warning labels

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Romer, PhD, Principal Investigator — University of Pennsylvania; Ellen Peters, PhD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Lazenby Hall, Ohio State University, Columbus, Ohio
  - Annenberg Public Policy Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Evans AT, Peters E, Strasser AA, Emery LF, Sheerin KM, Romer D. Graphic Warning Labels Elicit Affective and Thoughtful Responses from Smokers: Results of a Randomized Clinical Trial. PLoS One. 2015 Dec 16;10(12):e0142879. doi: 10.1371/journal.pone.0142879. eCollection 2015. PMID 26672982